CLINICAL TRIAL: NCT03665168
Title: A Multidimensional Strategy to Improve Quality of Life of Patients With Multiple Symptoms and Palliative Care Needs
Acronym: MuSt-PC
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: 201800366
Record Dates: First submitted 2018-09-07; First posted 2018-09-11 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Palliative Medicine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients in the palliative stage: Adult patients in various settings will be included (General Practioners practices, home care facilities, general and academic hospitals, hospices) and with any underlying life-limiting disease.

SUMMARY:
A nationwide, cross-sectional study, to determine the prevalence of symptoms of patients in the palliative phase in various care settings will be performed within a set period of two weeks in September 2018 and two weeks in November 2018. The participating settings will be selected by a total of seven coordinators, one for each consortium of palliative care in the Netherlands. To identify common combinations of symptoms and for multidimensional screening the Utrecht Symptom Diary-4 Dimensional (USD-4D) and Utrecht Symptom Diary (USD), a Dutch instrument based on the Edmonton Symptom Assessment Scale, will be used. The current protocol focuses on the cross-sectional study.

DETAILED DESCRIPTION:
The Utrecht Symptom Diary-4 dimensional (USD-4D), a Dutch instrument based on the Edmonton Symptom Assessment Scale, will be used for multidimensional screening and assessment of intensity and prevalence of symptoms. The questionnaire assesses twelve symptoms: pain, sleeping problems, dry mouth, dysphagia, anorexia, constipation, nausea, dyspnoea, fatigue, anxiety, depressed mood and confusion. This is measured on a numeric scale from 0 (no complaints) to 10 (worst imaginable or intolerable).

The prevalence of symptoms will be described by frequencies, dichotomizing symptom scores in absent (0 on NRS) or present (1 or higher on NRS). Symptom scores of 4 or higher on NRS are considered clinically relevant.

There is a possibility to add two more complaints not enlisted and to prioritise the problems which should be addressed first by the HCP.

Quality of life is assessed using a (un)well-being measure and the opportunity to score the experienced value of life.

Finally, five multidimensional questions will screen for mental capacity ("draagkracht"), the relationship with loved ones and thoughts concerning end of life. These multidimensional questions will be filled out together with the HCP. Therefore the HCP decides beforehand whether those questions will be asked.

The USD-4D will be filled out only once by participating patients without follow-up. The patients will be asked to fill out the following characteristics: age, gender, education level, cultural background, living situation, underlying disease, comorbidities, performance score, medication groups and interventions.

The estimated time to fill out both questionnaires is fifteen to twenty-five minutes.

ELIGIBILITY:
Patient selection will be performed by health care providers in the participating settings.

Inclusion Criterium:

• Patients of whom the health care professional answers "no" to the question "Would I be surprised if this patient died in the next 12 months ?".

Exclusion Criterium:

•Patients unable or unwilling to self-assess their symptoms

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients in various settings will be included (GP practices, home care facilities, general and academic hospitals, hospices) and with any underlying life-limiting disease
Sampling Method: Non-Probability Sample
Enrollment: 659 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of multiple, simultaneously occurring symptoms | 4 weeks
  Prevalence of multiple, simultaneously occurring symptoms (symptom clusters) in patients in the palliative phase in Dutch care settings (GP practices, home care facilities, general and academic hospitals, hospices).

SECONDARY OUTCOMES:
Prevalence of each separate symptom | 4 weeks
  For each symptom assessed (pain, sleeping problems, dry mouth, dysphagia, anorexia, constipation, nausea, dyspnoea, fatigue, anxiety, depressed mood and confusion) we will ask patients to score how they feel. In a Numerical Rating Scale (NRS), patients are asked to circle the number between 0 and 10 that fits best to their experienced intensity of complaints. Zero represents 'no complaint at all' whereas the upper limit represents 'the worst (pain, nausea, etc.) ever possible'.
Clinically relevant symptoms | 4 weeks
  For each symptom assessed (pain, sleeping problems, dry mouth, dysphagia, anorexia, constipation, nausea, dyspnoea, fatigue, anxiety, depressed mood and confusion) we will ask patients to score how they feel. In a Numerical Rating Scale (NRS), patients are asked to circle the number between 0 and 10 that fits best to their experienced intensity of complaints. Zero represents 'no complaint at all' whereas the upper limit represents 'the worst (pain, nausea, etc.) ever possible'. All scores of 4 and higher are considered clinically relevant.
Quality of life (single question with numeric rating scale) | 4 weeks
  Opportunity to score the experienced quality of life with the question: "how do you feel at this moment?". In a Numerical Rating Scale (NRS), patients are asked to circle the number between 0 and 10 that fits best to their wellbeing. Zero represents 'feeling very well' whereas the upper limit (10)represents 'feeling very bad'.
Symptom burden (multidimensional questions of Utrecht Symptom Diary-4Dimensional) | 4 weeks
  Five multidimensional theses will screen for mental capacity, the relationship with loved ones and thoughts concerning end of life. The following theses are presented:
  * I have the chance to be myself
  * I can bear what happens to me
  * I can let go of my loved ones
  * I am living a balanced life
  * Thoughts at the end of life gives me peace of mind
  In a Numerical Rating Scale (NRS), patients are asked to circle the number between 0 and 10 that fits best to their experienced feeling. Zero represents 'totally agree' whereas the upper limit represents 'totally disagree'. These values will be descriptive, a higher or lower value is not necessarily a better or worse outcome.
Symptoms per care setting | 4 weeks
  Number of participants with assessed complaints (pain, sleeping problems, dry mouth, dysphagia, anorexia, constipation, nausea, dyspnoea, fatigue, anxiety, depressed mood and confusion) per care setting (general practitioners practices, home care facilities, general and academic hospitals, hospices)
Symptoms per underlying disease | 4 weeks
  Number of participants with assessed complaints (pain, sleeping problems, dry mouth, dysphagia, anorexia, constipation, nausea, dyspnoea, fatigue, anxiety, depressed mood and confusion) per underlying disease (most probably incurable cancer, chronic obstructive pulmonary disease, heart failure and end-stage renal disease).

CONTACTS AND LOCATIONS:
Overall Officials: An KL Reyners, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands